CLINICAL TRIAL: NCT02440503
Title: Effect of Complementary Feeding With Different Macronutrient Quantities on Growth and Body Composition: a Follow-up Trial
Brief Title: How Infant Diets Would Affect Growth in Early Childhood
Acronym: FYI-FU
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0489; UL1TR001082 (NIH)
Record Dates: First submitted 2014-06-25; First posted 2015-05-12 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Growth; Body Composition; Gut Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — stool samples will be collected for microbiome analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators research group conducted a feeding study in 2012 (IRB 07-0003) that included breastfed infants consuming different infant solid foods. The investigators results showed that different solid foods, especially the protein content of the food, is important on infant's gut bacteria profile and growth. Although the first year of life is critical in obesity development later in life, data are very limited on the effect of protein from solid foods, an important component of infant diet, especially in breast-fed infants. In this study, the investigators will re-contact these participants, who are now in their early childhood (~5 years old), to evaluate the long-term effect of various macronutrient quantities in solid foods, by assessing the participants' growth, body composition, and gut bacteria profile.

ELIGIBILITY:
Inclusion Criteria:

* Those participants who completed the initial trial when they were infants.

Exclusion Criteria:

* None

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 4-6 years of age
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Age adjusted height | Day 1: one time assessment during the participant's visit to Colorado Children's hospital
  observational, one time assessment. The hospital visit is scheduled according to the participant's availability.
Age adjusted weight | Day 1: one time assessment during the participant's visit to Colorado Children's hospital
  observational, one time assessment. The hospital visit is scheduled according to the participant's availability.

SECONDARY OUTCOMES:
Percent body fat | Day 1: one time assessment during the participant's visit to Colorado Children's hospital
  Body composition using DEXA scan will be assessed during the hospital visit

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Tang, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UC Denver, Aurora, Colorado, United States